CLINICAL TRIAL: NCT05779852
Title: Pain Management of Amputation Wounds With AutoHypnosis
Acronym: MODOUPAAH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 35RC20_8896_MODOUPAAH; 2022-A00638-35 (Other: N°ID-RCB)
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-06

CONDITIONS: Vascular Surgical Procedures
Keywords: lower extremity artery disease; self-hypnosis; amputation care
MeSH Terms: interventions — Hypnosis; Bandages

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-hypnosis and care (Experimental)
  Interventions: Other: self-hypnosis and dressing
- care (Other)
  Interventions: Other: dressing

INTERVENTIONS:
Other: self-hypnosis and dressing — self-hypnosis during dressing
  Arms: self-hypnosis and care
Other: dressing — dressing without self-hypnosis
  Arms: care

SUMMARY:
Amputation in vascular surgery mainly concerns the lower limb and is often linked to Obliterative Arterial Disease of the Lower Limbs. It indicates the impossibility or failure of revascularisation after an exhaustive assessment aimed at saving the limb. It is also performed to limit the spread of gangrene, an affection of the limb that can evolve into septicaemia. The principle is to amputate in a healthy and vascularised area to allow good healing of the amputation stump.

Amputations of one, several or all toes, called complete transmetatarsal amputations, may take several months to heal. Amputations require directed healing and, above all, monitoring of the underlying tissues of the amputated area by daily detersions and wiping performed by a nurse at home. The mechanical detersion of the wound necessary for the healing process and cell migration, as well as optimal deep meshing, facilitate the evolution of the healing process.

These treatments often cause pain, despite oral analgesics and local anaesthetics prior to the treatment.

For several years, studies have shown the benefits of hypnosis in modifying the perception of pain, particularly during treatment.

Studies have also shown that self-hypnosis allows a reduction in the intensity of pain.

The clinical experience of the vascular surgery department of the University Hospital of Rennes suggests that patients who use self-hypnosis during the daily dressing of their amputation experience the moment more serenely, increasing their comfort and decreasing their pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Naïve to amputation procedures;
* Amputated, within 24 hours prior to inclusion, one, more or all toes
* Pain level on the Numerical Scale ≥ 3 during the first dressing;
* Affiliated to a social security scheme;
* Having signed a free, informed and written consent.

Exclusion Criteria:

* Cognitive impairments that limit understanding of instructions;
* Cultural limitations reducing abstraction skills;
* Previous practice of hypnosis;
* Contraindications to hypnosis: Bipolar disorder or decompensated schizophrenia;
* Chronic non-vascular pain;
* Already in care for painful chronic wounds (ulcer wounds, bedsores...)
* On morphine before surgery;
* Analgesia by perineural catheter;
* Protected person (adult subject to legal protection (safeguard of justice, curatorship, guardianship), person deprived of liberty, pregnant woman (declarative), nursing woman and minor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Level of pain | Day 2 (during the 3rd post-operative amputation bandage)
  pain self-assessment numerical scale graduated from "0" - no pain - to "10" - unimaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Claudie BOUFFORT, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France